CLINICAL TRIAL: NCT06254404
Title: Impact of Protamine Dose Reduction on Platelet Aggregation After Extracorporeal Circulation for Minimally Invasive Aortic Valve Replacement Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Benjamin Javillier, MD, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LowProt
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Protamine Dose; Protamine Adverse Reaction
MeSH Terms: interventions — Protamines

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose of Protamine (Active Comparator)
  Interventions: Drug: Low dose protamine
- Normal dose of protamine (Experimental)
  Interventions: Drug: Low dose protamine

INTERVENTIONS:
Drug: Low dose protamine — Administration of 70% of the normal dose of protamine

SUMMARY:
Determining the minimum effective dose of protamine after extracorporeal circulation for mini-sternotomy aortic valve replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Mini-sternotomy aortic valve replacement surgery
* Major patients

Exclusion Criteria:

* Hypersensitivity to protamine
* Coagulation Abnormalities
* Heparin allergy
* Pregnant women
* Jehovah's Witnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Minimum effective dose of protamine after extracorporeal circulation. A bottom-up and top-down method will define CP 50. | 24 hours